CLINICAL TRIAL: NCT02139423
Title: Feasibility to Achieve, Before One Month of Age, the Diagnosis of Congenital CMV Diagnosis and the Formal Audiologic Assessment in Newborns Who Failed Newborn Hearing Screening
Brief Title: Diagnosis of Congenital CMV Infection in Neonates Who Failed Newborn Hearing Screening
Acronym: CymeAudit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRC12025
Record Dates: First submitted 2014-04-28; First posted 2014-05-15 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Congenital Cytomegalovirus Infection
Keywords: Congenital cytomegalovirus infection; newborn universal hearing screening
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All newborns who fail universal newborn (Experimental): CMV PCR
  Interventions: Other: CMV PCR

INTERVENTIONS:
Other: CMV PCR
  Other Names: CMV PCR results are communicated to the relevant clinicians in real time.

SUMMARY:
Universal hearing screening at birth by use of otoacoustic emission (OAE) is now offered in most maternities in France to detect symptomatic hearing impairment at birth but screening of cCMV infection is not coupled with this screening. In this study, the feasibility of achieving before one month of age the diagnosis of congenital CMV diagnosis and as well as the confirmation of hearing loss in newborns who failed newborn hearing screening will be tested.

DETAILED DESCRIPTION:
Congenital cytomegalovirus (cCMV) is the most frequent congenital infection in France. Around 90% of cCMV infected infants are asymptomatic at birth, of whom 7 to 20% develop sensorineural hearing loss (SNHL). cCMV explains at least 10% of all hearing loss cases in young children. Early antiviral treatment (implemented before 1 month of age) with ganciclovir or valganciclovir can improve hearing outcome. In the absence of universal screening, cCMV remains largely undetected because most infected neonates are asymptomatic or have non-specific symptoms. When symptoms become apparent or develop, it may be too late for confirmation that the infection is of congenital origin becausediagnosis of congenital infection is based on the detection of CMV in samples collected within 2 to 3 weeks after birth. The presence of CMV in samples collected after this time may represent postnatal infection which does not carry the risk of hearing loss or neurodevelopmental sequelae. Universal hearing screening at birth by use of otoacoustic emission (OAE) is now offered in most maternities in France to detect symptomatic hearing impairment at birth but screening of cCMV infection is not coupled with this screening. In this study, the feasibility of achieving before one month of age the diagnosis of congenital CMV diagnosis and as well as the confirmation of hearing loss in newborns who failed newborn hearing screening will be tested.

ELIGIBILITY:
Inclusion Criteria:

* All newborns who have failed universal newborn screening

Exclusion Criteria:

* Neonates whose mothers would object to the use of their child's medical data

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 235 (Actual)
Dates: Start 2014-11-22 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Number of days necessary to obtain the result of cCMV infection diagnosis and the audiological result after formal assessment | 1 month

SECONDARY OUTCOMES:
Measurement of CMV by quantitative PCR | 4 months
  correlation between the results obtained from saliva and from blood (isolated from Guthrie cards)
Number of children for whom the result of the formal audiological assessment has been obtained | 4 months
Number of children with cCMV infection and confirmed hearing loss in whom antiviral therapy has been initiated within the first month of life | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Leruez-Ville, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker-Enfants-Malades, Paris, France

REFERENCES:
- [Derived] Fourgeaud J, Boithias C, Walter-Nicolet E, Kermorvant E, Couderc S, Parat S, Pol C, Mousset C, Bussieres L, Guilleminot T, Ville Y, Nkam L, Grimaldi L, Parodi M, Leruez-Ville M. Performance of Targeted Congenital Cytomegalovirus Screening in Newborns Failing Universal Hearing Screening: A Multicenter Study. Pediatr Infect Dis J. 2022 Jun 1;41(6):478-481. doi: 10.1097/INF.0000000000003474. Epub 2022 Jan 27. PMID 35093998